CLINICAL TRIAL: NCT03881436
Title: Assessment of MRI Tractography for Pelvic Floor Sphincter Analysis
Acronym: TractoCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-005
Record Dates: First submitted 2019-03-04; First posted 2019-03-19 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Inflammatory Bowel Disease; Neoplastic Pathology
Keywords: Anatomy; Fiber tractography; Pelvic floor; Diffusion Tensor Imaging (DTI); Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic MRI (Experimental): This arm involves patients undergoing a pelvic MRI.
  At the end of the planned sequence, but before any contrast agent injection:
  * Acquisition of a an additional anatomical T2 SPACE sequence
  * Acquisition of a tractography Diffusion Tensor Imaging (DTI) sequence All acquisitions will be done in an acceptable duration (less than 45 minutes)
  Interventions: Diagnostic Test: MRI with DTI sequence
- Pelvic surgery (Experimental): This arm involves patients undergoing a pelvic surgery and coming for a postoperative MRI. An additional MRI is performed before the surgery and additional sequences are added to the planned postoperative MRI, at the end of the planned sequence, but before any contrast agent injection:
  * Acquisition of a an additional anatomical T2 SPACE sequence
  * Acquisition of a tractography Diffusion Tensor Imaging (DTI) sequence All acquisitions will be done in an acceptable duration (less than 45 minutes)
  Interventions: Diagnostic Test: MRI with DTI sequence

INTERVENTIONS:
Diagnostic Test: MRI with DTI sequence — At the end of the planned sequence, but before any contrast agent injection:
  * Acquisition of a an additional anatomical T2 SPACE sequence
  * Acquisition of a tractography DTI sequence

SUMMARY:
Urinary and faecal incontinences generally come from a dysfunction of the pelvic floor muscles, and more particularly the sphincters. Among other causes, they may be related to accidental trauma, obstetric or iatrogenic. On this last point, the incidence of surgical interventions on the bladder collar and on the anal canal on the prevalence of incontinences can be underlined.

MRI tractography could be an interesting tool to visualize in 3D the structure of pelvic sphincters and their lesions. It may thereby establish the link with observed dysfunctions, thus potentially providing a complement to the urological and proctographic examinations already carried out.

The objective of this study is, first, to define the sensitivity of the MRI tractography for the visualization of the pelvic sphincters architecture regardless of the gender. In a second time, it will give a description of normal and abnormal (pathological cases) tractography, as well as a descriptive post-surgery. The other interest of this study is the assessment of the information provided by pelvic sphincters tractography on a panel of various and frequently encountered situations in clinical routine at the IHU.

DETAILED DESCRIPTION:
Urinary and faecal incontinences are psychologically difficult to live with. These disorders generally come from a dysfunction of the pelvic floor muscles, and more particularly the sphincters: the urethral sphincter at the level of the urinary tract, and the anal sphincter at the level of the defecatory apparatus. The causes leading to urinary or faecal incontinence are multiple. They may be related to age or weight, or to accidental trauma, obstetric or iatrogenic. On this last point, the incidence of surgical interventions on the bladder collar and on the anal canal on the prevalence of incontinences can be underlined.

In case of dysfunction, the sphincters can be scanned by imaging, including MRI, to assess the thickness or detect the presence of scars. The current MRI examinations in clinical routine are not capable to characterize the complex architecture of these muscles. MRI tractography, mainly known as a tool for visualisation and characterisation of white matter fibers in the brain via the acquisition of DTI (Diffusion Tensor Imaging) sequences, could be an interesting tool to visualize in 3D the structure of pelvic sphincters and their lesions. It may thereby establish the link with observed dysfunctions, thus potentially providing a complement to the urological and proctographic examinations already carried out.

Some studies have already shown that MRI is an ideal method for visualizing pelvic floor muscle fibers in women. As far as it is known, there are no studies in the literature on pelvic sphincter tractography. The objective is, first, to define from this initial study the sensitivity of the method for the visualization of the pelvic sphincters architecture regardless of the gender. In a second time, it will give a description of normal and abnormal (pathological cases) tractography, as well as a descriptive post-surgery. The results found in each of these situations can be compared in order to evaluate the sensitivity and contribution of MRI tractography for the diagnosis of pelvic sphincter dysfunctions and their management, as well as to evaluate the impact of surgery.

The other interest of this study is the inclusion of both patients consulting for a simple diagnosis and those coming for a pre- and post-operative examination. This will allow the assessment of the information provided by pelvic sphincters tractography on a panel of various and frequently encountered situations in clinical routine at the IHU.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 18 years old
2. Patient able to receive and understand information related to the study and give written informed consent
3. Patient affiliated to the French social security system
4. Patient undergoing a pelvic MRI examination whose result at the end of the T2 sequences in the 3 section planes shows the absence of pathology or a distant pathology that does not affect the pelvic sphincters OR Patient undergoing a pelvic surgery including fistula treatment, abscess treatment, sigmoid mucosectomy or rectal mucosectomy

Exclusion Criteria:

1. Patient who previously had a therapeutic procedure affecting the sphincters
2. Patient with hip prostheses
3. Patient with contraindications to MRI:

   * pacemaker or automatic defibrillator, pump
   * implanted
   * auditory, anal, painkiller neurostimulator, etc ...
   * ferromagnetic bodies in soft tissues, body
   * intraocular foreigners, cerebrovascular clips
   * claustrophobia
4. Patient presenting, in the judgment of the investigator, an illness that may prevent participation in the procedures provided by the study
5. Pregnant or lactating patient
6. Patient in exclusion period (determined by a previous or a current study)
7. Patient under guardianship or trusteeship
8. Patient under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
The ability of MRI tractography to visualize the muscular architecture of pelvic sphincters evaluated with a Likert score. | 1 day for the "Pelvic MRI" group - 2 months for the "Pelvic surgery" group
  This criterion is quantitative and is evaluated on the basis of a Likert score varying between 1 and 5 which will be attributed to each sphincter.
  * Score 1 = no reconstruction: sphincter not visualised
  * Score 2 = insufficient reconstruction: the fiber architecture is incoherent and / or few fibers are rebuilt
  * Score 3 = acceptable reconstruction: the reconstructed fibers provide an overview of sphincter architecture despite the presence of incoherent or missing fibers
  * Score 4 = satisfactory reconstruction: the sphincter is generally well reconstructed, little incoherence and missing fibers
  * Score 5 = excellent reconstruction: the appearance of the sphincter reflects the expected anatomy, without missing or inconsistent fibers.

SECONDARY OUTCOMES:
Evaluation of the sphincter orientation based on a color gradient. | 1 day for the "Pelvic MRI" group - 2 months for the "Pelvic surgery" group
  The reconstruction of the muscle fibers in tractography is done according to a precise color code (blue if orientation up-down, green for front-back, and red for left-right).
  The analysis will be done on the color gradient.
Thickness of the sphincters evaluated in millimetres | 1 day for the "Pelvic MRI" group - 2 months for the "Pelvic surgery" group
  The thickness of the sphincters will be measured in millimetres
Fractional Anisotropy (FA) Values in Sphincter Fibres | 1 day for the "Pelvic MRI" group - 2 months for the "Pelvic surgery" group
  Fractional anisotropy (FA) is a scalar value between zero and one that describes the degree of anisotropy of a diffusion process. A value of zero means that diffusion is isotropic, i.e. it is unrestricted (or equally restricted) in all directions. A value of one means that diffusion occurs only along one axis and is fully restricted along all other directions.
Apparent Diffusion Coefficient (ADC) Values in Sphincter Fibres | 1 day for the "Pelvic MRI" group - 2 months for the "Pelvic surgery" group
  Apparent diffusion coefficient (ADC) is a measure of the magnitude of diffusion (of water molecules) expressed in units of square millimetres per second (mm2/s).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine ROY, MD, Principal Investigator — Service de Radiologie et d'Echographie, NHC Strasbourg
Locations (1):
- Service de Radiologie et d'Echographie, NHC Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zijta FM, Froeling M, van der Paardt MP, Lakeman MM, Bipat S, van Swijndregt AD, Strijkers GJ, Nederveen AJ, Stoker J. Feasibility of diffusion tensor imaging (DTI) with fibre tractography of the normal female pelvic floor. Eur Radiol. 2011 Jun;21(6):1243-9. doi: 10.1007/s00330-010-2044-8. Epub 2011 Jan 1. PMID 21197534
- [Background] Zijta FM, Lakeman MM, Froeling M, van der Paardt MP, Borstlap CS, Bipat S, Montauban van Swijndregt AD, Strijkers GJ, Roovers JP, Nederveen AJ, Stoker J. Evaluation of the female pelvic floor in pelvic organ prolapse using 3.0-Tesla diffusion tensor imaging and fibre tractography. Eur Radiol. 2012 Dec;22(12):2806-13. doi: 10.1007/s00330-012-2548-5. Epub 2012 Jul 14. PMID 22797954
- [Background] Rousset P, Delmas V, Buy JN, Rahmouni A, Vadrot D, Deux JF. In vivo visualization of the levator ani muscle subdivisions using MR fiber tractography with diffusion tensor imaging. J Anat. 2012 Sep;221(3):221-8. doi: 10.1111/j.1469-7580.2012.01538.x. Epub 2012 Jul 4. PMID 22757638